CLINICAL TRIAL: NCT07058051
Title: Cross-sectional Study to Characterize Real World Burden of Disease in Patients With Vitiligo in China
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H25-976
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non-Segmental Vitiligo

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate the patterns of treatment, healthcare resources utilized and the burdens associated with non-segmental vitiligo (NSV) amongst participants in China

This study is a cross-sectional, multicenter, observational study of vitiligo patients in China. The cross-sectional design is sufficient to characterize the overall current burden of NSV.

DETAILED DESCRIPTION:
Cross-Sectional

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age ≥ 12.
* Chinese patients meet the diagnosis of Non-Segmental Vitiligo (NSV) and 5≤ Total Vitiligo Area Scoring Index (T-VASI<50) with or without facial involvement.
* Medical history available within the last 6 months.
* Ability to understand the questionnaires, with parental support as required for adolescents (between ≥ 12 and < 18 years of age at inclusion visit).
* Willing to provide a patient authorization form to use and disclose personal health information (or informed consent, where applicable) to participate in the study; for adolescent subjects, authorization and/or consent will be provided by a parent or legal guardian, where applicable.

Exclusion Criteria:

* Unable or unwilling to comply with study requirements and electronic Patient-Reported Outcome (ePRO) collection.
* Segmental or localized vitiligo.
* Greater than 33% leukotrichia in areas of vitiligo on the face or on the body.
* History of active skin disease other than vitiligo that could interfere with the assessment of vitiligo.
* Patients who are participating in interventional clinical trial(s) at time of study visit.
* Patients who are currently receiving treatment with any investigational drug/device/intervention or have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) prior to enrollment.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese patients with non-segmental vitiligo and 5≤T-VASI<50 will be included. The NSV patients will be consecutively enrolled via convenience sampling in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-07-17 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Total Vitiligo Area Scoring Index (T-VASI) | At Inclusion Visit (Day 1)
  The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100, with higher scores indicating more severe disease.
Vitiligo Quality of Life Scale (VitiQoL) | At Inclusion Visit (Day 1)
  The VitiQoL is an 16-item instrument assessing impact of vitiligo on quality of life. 15 items are scored on a 7-point Likert scale, ranging from "not at all" to "all the time". An additional item (not contributing to total score) assesses current severity of condition on a 7-point scale ranging from "no skin involvement" to "most severe case"

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- China (4):
  - Dermatology Hospital of Southern Medical University /ID# 276921, Guangzhou, Guangdong
  - Wuhan Integrated TCM & Western Medicine Hospital（Wuhan No.1 Hospital) /ID# 276919, Wuhan, Hubei
  - Suzhou Municipal Hospital /ID# 276948, Suzhou, Jiangsu
  - Shandong Dermatological Hospital /ID# 276918, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=H25-976